CLINICAL TRIAL: NCT04886921
Title: Post-mastectomy Women Underwent Transverse Rectus Abdominis Musculocutaneous Flap (TRAM) Surgery: Its Influence on Abdominal Muscle Function and the Effects of Therapeutic Exercises
Brief Title: Women Underwent TRAM Surgery: Its Influence on Abdominal Muscle Function and the Effects of Therapeutic Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KMUH-IRB-970469
Record Dates: First submitted 2021-05-11; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-02

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TRAM abdominal muscle training group (Experimental): Patients were recruited at least 6 months after the muscle-sparing (MS) pedicled Transverse rectus abdominis musculocutaneous (TRAM) flap procedure and at least 1 month after the conclusion of the last chemotherapy course, if any.
  All subjects will receive 1-hr training sessions consisting of core stability exercises for 12 weeks for the TRAM group.
  Interventions: Behavioral: Abdominal muscle training
- TRAM control group (No Intervention): Patients were recruited at least 6 months after the muscle-sparing (MS) pedicled Transverse rectus abdominis musculocutaneous (TRAM) flap procedure and at least 1 month after the conclusion of the last chemotherapy course, if any.
  The control group was not received any exercise program.
- Healthy women group (No Intervention): A control group comprising female volunteers who were apparently healthy and had comparable socioeconomic backgrounds and physical conditions was recruited by convenience sampling from communities.

INTERVENTIONS:
Behavioral: Abdominal muscle training — Participants will receive 12-week, 60 minutes, 36-session abdominal muscle training in the TRAM women. Aimed to evaluate the effects on abdominal muscle functions after 12 weeks abdominal muscle training in the TRAM women. Outcome measures were the clinical tests for trunk muscle strength, endurance and one-leg standing was also used to exam the abdominal muscle function.
  Arms: TRAM abdominal muscle training group

SUMMARY:
The unilateral transverse rectus abdominis musculocutaneous (TRAM) flap is a major operation widely used for breast reconstruction. It is hypothesized that this surgery has the potential risk of weakening the abdominal wall because it disrupts the integrity of the rectus abdominis muscle (RA), therefore, alters the insertion of the oblique muscles and the biomechanical relationship between the RA muscle and adjacent structures. The purposes of this study were to examine the effects of the TRAM flap surgery on muscle size of abdominal muscles, strength and endurance of trunk muscles, strength and endurance of core stability, as well as the effects of therapeutic exercises on it in post-mastectomy women underwent TRAM surgery.

DETAILED DESCRIPTION:
This first year of the proposed study was aimed to understand the impacts on abdominal muscle functions. We design a case-control, cross-sectional study. There were 46 women who have undergone TRAM flap and 36 age-matched healthy women. We recorded the biomechanic and electromyographic responses during voluntary limb movements and elicited by unexpected support surface translations and tilts in standing. A six-camera Qualisys motion system was used. Ground reaction forces and moments were acquired by one Kisler force plate. Surface electromyography electrodes were used to record the activity of selected trunk and limb muscles. The second year was aimed to evaluate the effects on abdominal muscle functions after 12 weeks abdominal muscle training in the TRAM women. Outcome measures were the clinical tests for trunk muscle strength, endurance and one-leg standing was also used to exam the abdominal muscle function.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults

   * Their age should be ranged between 30 - 60 years
2. TRAM flap surgery patients

   * at least 6 months after the MS pedicled TRAM flap surgery

Exclusion Criteria:

1. Healthy adults

   * a history of injury resulting in an inability to perform activities of daily living
   * scoliosis or spinal surgery
   * neurological, neuromuscular, rheumatological or systemic diseases
2. TRAM flap surgery patients

   * tumor distant metastasis
   * a history of injury resulting in an inability to perform activities of daily living
   * scoliosis or spinal surgery
   * neurological, neuromuscular, rheumatological or systemic diseases

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2009-02-24 (Actual); Primary Completion 2014-09-08 (Actual); Study Completion 2014-09-08 (Actual)

PRIMARY OUTCOMES:
Changes in thickness of abdominal wall muscles at 12-week | The assessments will be conducted 1 and 12 weeks following the intervention
  Using the Ultrasound imaging to measure the thickness of all abdominal wall muscles at rest and in an isometric contraction.
Changes in the cross-sectional area of the rectus abdominis muscle (RA) muscle at 12-week | The assessments will be conducted 1 and 12 weeks following the intervention
  Using the Ultrasound imaging to measure the cross-sectional area of the rectus abdominis muscle at rest and in an isometric contraction.
Changes in strength of the trunk muscles at 12-week | The assessments will be conducted 1 and 12 weeks following the intervention
  Using the dynamometer and clinical tests (prone extension, curl-up and rotational curl-up) to measure the trunk strength
Changes in endurance of the trunk muscles at 12-week | The assessments will be conducted 1 and 12 weeks following the intervention
  Using the clinical tests (abdominal muscle test for strength, unsupported double bend leg lifting for static endurance) to measure the endurance of trunk muscles
Changes in balanced functions at 12-week | The assessments will be conducted 1 and 12 weeks following the intervention
  Using the seconds in the following static position to measure the balance: one-leg standing with the other lift-leg 1 inch of ground clearance; single leg standing with the other lift-leg hip flexion 90 degrees and the tibia vertical to the floor.
Changes in muscle activity of selected trunk and limb muscles at 12-week | The assessments will be conducted 1 and 12 weeks following the intervention
  Using A six-camera Qualisys motion system to measure the muscle activity of selected trunk and limb muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jiun Liaw, Study Director — Kaohsiung Medical University Department of Physical Therapy Associate Professor

IPD SHARING:
Plan to Share IPD: No
Currently in the submission stage ,and then share with other researchers after publication